CLINICAL TRIAL: NCT01912040
Title: A Prospective, Open Label, Single Arm Cohort Study to Assess the Frequency of Adverse Reactions of Locally Manufactured 123I-metaiodobenzylguanidine in Routine Clinical Use
Brief Title: Study Of the Safety of Locally Manufactured 123I-metaiodobenzylguanidine(MIBG) in Routine Clinical Use
Status: Withdrawn | Type: Observational
Why Stopped: Issues with obtaining precursor materials for synthesis
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: 123Iodine MIBG
Record Dates: First submitted 2013-07-12; First posted 2013-07-30 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2013-07

CONDITIONS: Adrenergic Pathology
Keywords: Safety profile; locally produced 123 Iodine MIBG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Administration of 123Iodine MIBG to the patients referred .
  Interventions: Drug: Administration of 123Iodine MIBG

INTERVENTIONS:
Drug: Administration of 123Iodine MIBG — Patients will be administered the locally produced 123 Iodine MIBG
  Other Names: None applicable

SUMMARY:
Assessing 123 Iodine MIBG produced locally for safety while being used in clinical practice to help in patient management decisions.

DETAILED DESCRIPTION:
We will be assessing for adverse reactions of patients injected with locally manufactured 123 Iodine MIBG. With monitoring of blood pressure and heart rate following injection and any potential immediate side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with potential Adrenergic pathology

Exclusion Criteria:

* Pregnant or breast feeding females
* Hypersensitivity to MIBG

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Those patients referred for MIBG assessment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Safety profile of the 123Iodine MIBG | BP and Heart rate for 24 hours after injection.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ross, MD, Principal Investigator — Division Head, Nuclear Medicine
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada